CLINICAL TRIAL: NCT03471481
Title: Magnesium as a Mediator of Bone and Vitamin D Metabolism in Patients on Antiepileptic Drug Therapy
Status: Terminated | Type: Observational
Why Stopped: Closure of Drexel University Hahnemann Hospital where Referring Physician Worked
Sponsor: Drexel University (Other)
Responsible Party: Sponsor
Other Study IDs: 150003722
Record Dates: First submitted 2018-03-14; First posted 2018-03-20 (Actual); Last update posted 2021-03-01 (Actual); Status verified 2019-11

CONDITIONS: Epilepsy; Magnesium Deficiency; Vitamin D Deficiency
MeSH Terms: conditions — Epilepsy; Magnesium Deficiency; Vitamin D Deficiency

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Serum and urine samples
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: No Intervention. Study is Cross Sectional in nature — No Intervention. Study is cross sectional in nature

SUMMARY:
The objective of this study is to determine the role of magnesium on bone and vitamin D metabolism in patients receiving anti-epileptic medications.

ELIGIBILITY:
Inclusion Criteria:

* Individuals receiving anti-epileptic drugs as a treatment for epilepsy

Exclusion Criteria:

* Individuals who are pregnant or breastfeeding, receiving cancer treatments, have liver or kidney diseases, autoimmune diseases, or other diseases that may interfere with vitamin D and magnesium metabolism.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Individuals diagnosed with epilepsy and on medications
Sampling Method: Non-Probability Sample
Enrollment: 7 (Actual)
Dates: Start 2015-08-10 (Actual); Primary Completion 2019-08-01 (Actual); Study Completion 2019-08-01 (Actual)

PRIMARY OUTCOMES:
Bone mineral density | 1 time point - baseline
  Will be measured at Tibia, Hip and Total Body using a DXA scan

SECONDARY OUTCOMES:
Ionized Magnesium in serum | 1 time point - baseline
  This will be assayed in the serum
Vitamin D - 25 hydroxy vitamin D | 1 time point - baseline
  This will be assayed in the serum

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Drexel University Nutrition Sciences Research Lab, Philadelphia, Pennsylvania
  - Drexel University, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: Undecided